CLINICAL TRIAL: NCT00864955
Title: Damage to DNA Caused by UV-A Irradiation: Photochemical Mechanism and Cutaneous Parameters Involved in the Formation of Cyclobutane Pyrimidine Dimers
Brief Title: Cutaneous DNA Damage Caused by UV-A Irradiation
Acronym: DIMUVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government)
Responsible Party: Direction de la Recherche Clinique, University Hospital Grenoble
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DCIC 08 13
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Healthy Volunteers
Keywords: UV-A irradiation; Cyclobutane-Pyrimidine Dimer; Oxidative lesions; cutaneous phototype; UV-B irradiation; DNA damages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- phototype 2 (Experimental): Volunteers with cutaneous phototype 2
  Interventions: Radiation: UVA and UVB irradiation
- phototype 4 (Experimental): Volunteers with cutaneous phototype 4
  Interventions: Radiation: UVA and UVB irradiation

INTERVENTIONS:
Radiation: UVA and UVB irradiation — * 4 cutaneous biopsies for Ex-vivo irradiation
  * Determination of the minimal erythemic dose of UVA and UVB for each volunteer

SUMMARY:
The DIMUVA study aims to evaluate the correlation between cutaneous phototype and the nature and quantity of damage caused to cutaneous DNA after exposure to UV-A radiation.

DETAILED DESCRIPTION:
Due to their capacity to damage Deoxyribonucleic acid (DNA), Ultra-Violet (UV) radiation is one of the causes of skin cancers.

Until recently, the genotoxic effects of UV-A radiation, were poorly identified, in particular their capacity to lead to the dimerization of pyrimidine bases .

It is well known that the response to UV-A and UV-B radiations is different depending on the cutaneous phototype.

Thus, the aim of this study is to determine the correlation between cutaneous phototype and the quantity and nature (CPD or oxidative lesions) of damage caused to cutaneous DNA after an ex-vivo exposure to UV-A and UV-B radiations.

ELIGIBILITY:
Inclusion Criteria:

* Male,
* Between 18 and 35 years old,
* Healthy volunteers,
* Cutaneous phototype 2 or 4 according to the Fitzpatrick classification,
* Affiliation to the French Social Security.

Exclusion Criteria:

* History of photosensibility,
* Active smoking or stopped since less than one year,
* Dermatological pathology or treatment contra-indicating cutaneous irradiation and skin biopsies,
* Any chronic pathology susceptible to interfere with the evaluations related to the protocol,
* Allergy to local anaesthetics,
* Volunteers who take drugs and/or food complements acting on oxidative stress in the 8 weeks preceding inclusion,
* Volunteers who have take paracetamol or aspirin within 7 days prior to the inclusion visit,
* Subject in exclusion period for another biomedical research study,
* Subject having exceeded the threshold of annual compensation for biomedical research.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Phototype determination according to the Fitzpatrick classification Number of CPD and oxidative lesions determinated by the analysis of DNA from the skin biopsies after their ex-vivo exposure to UV-A - The CPD / Oxidative lesions ratio | Day 0

SECONDARY OUTCOMES:
Number of CPD and oxidative lesions determinated by the analysis of DNA from the skin biopsies after their exposure ex-vivo to UV-B. | Day 0
UV-A radiation exposure: Minimal erythemic dose - Number of CPD and oxidative lesions - CPD / oxidative lesions ratio | Day x
UV-B radiation exposure: Minimal erythemic dose - Number of CPD and oxidative lesions - CPD/oxidative lesions ratio | Day 0
antioxidant status and quantity of CPD, oxidative lesions after exposure to UV-A and UV-B radiations | day 2

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude BEANI, Pr, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - Centre d'investigation Clinique ,University Hospital Grenoble, Grenoble
  - Department of Dermatology, University Hospital Grenoble, Grenoble

REFERENCES:
- [Background] Brash DE. Sunlight and the onset of skin cancer. Trends Genet. 1997 Oct;13(10):410-4. doi: 10.1016/s0168-9525(97)01246-8. PMID 9351343
- [Background] Melnikova VO, Ananthaswamy HN. Cellular and molecular events leading to the development of skin cancer. Mutat Res. 2005 Apr 1;571(1-2):91-106. doi: 10.1016/j.mrfmmm.2004.11.015. PMID 15748641
- [Background] Cadet J, Sage E, Douki T. Ultraviolet radiation-mediated damage to cellular DNA. Mutat Res. 2005 Apr 1;571(1-2):3-17. doi: 10.1016/j.mrfmmm.2004.09.012. Epub 2005 Jan 26. PMID 15748634
- [Background] Douki T, Reynaud-Angelin A, Cadet J, Sage E. Bipyrimidine photoproducts rather than oxidative lesions are the main type of DNA damage involved in the genotoxic effect of solar UVA radiation. Biochemistry. 2003 Aug 5;42(30):9221-6. doi: 10.1021/bi034593c. PMID 12885257
- [Background] Dumaz N, Drougard C, Sarasin A, Daya-Grosjean L. Specific UV-induced mutation spectrum in the p53 gene of skin tumors from DNA-repair-deficient xeroderma pigmentosum patients. Proc Natl Acad Sci U S A. 1993 Nov 15;90(22):10529-33. doi: 10.1073/pnas.90.22.10529. PMID 8248141